CLINICAL TRIAL: NCT01906216
Title: Sorafenib With or Without Transarterial Chemoembolization (TACE) in Advanced Hepatocellular Carcinoma : A Multicenter, Randomized, Controlled Trial
Brief Title: Sorafenib Chemoembolization Evaluation Controlled Trial
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHDD-001
Record Dates: First submitted 2013-05-29; First posted 2013-07-24 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; sorafenib; transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib (Active Comparator): All subjects will take two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening). Sorafenib may be taken either with a low/moderate fat meal or without food. Subjects are to continue sorafenib according to the study protocol if the adverse events could be safely controlled.
  Interventions: Drug: Sorafenib
- Sorafenib combined with TACE (Experimental): Sorafenib will be supplied as 200 mg tablets. All subjects will take two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening). In addition, the subjects in this arm will receive the treatment of conventional transarterial chemoembolization. In all cases, TACE consists of an injection containing a mixture of chemotherapeutic agents(doxorubicin) and lipiodol followed by embolization with polyvinyl alcohol (PVA) or beads.
  Interventions: Drug: Sorafenib; Procedure: TACE

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be supplied as 200 mg tablets. All subjects will take two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening).
  Other Names: Bay 43-9006, Sorafenib (Nexavar®)
Procedure: TACE — The first treatment of TACE should be completed within 3-7 days after the administration of sorafenib started. In all cases, TACE consists of an injection containing a mixture of chemotherapeutic agents and lipiodol followed by embolization with polyvinyl alcohol (PVA) or beads until complete stasis was achieved in the tumor-feeding vessels.Tumor-feeding vessels should be selected/superselected whenever possible. TACE will be repeated "on demand" depending on the radiological response.
  Arms: Sorafenib combined with TACE

SUMMARY:
This prospective, multicenter, randomized, controlled study aims to evaluate the efficacy and safety of sorafenib combined with transarterial chemoembolization (TACE) in advanced hepatocellular carcinoma (HCC) patients compared with sorafenib alone, and to determine the prognostic factors that influence the survival.

Data on the efficacy and safety of sorafenib in combination with TACE in patients with advanced HCC are lacking. Because in western countries, advanced HCC is considered as a contraindication for TACE treatment. However, clinical practice patterns differ markedly between Asia and western countries: in Asia TACE is performed in selected advanced HCC patients. We consider sorafenib combined with TACE could achieve better survival benefit than sorafenib alone in selected advanced HCC patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To compare the overall survival of selected advanced HCC patients treated with sorafenib combined with TACE with sorafenib alone.

SECONDARY OBJECTIVES:

1. To compare the time to progression (TTP, according to mRECIST criteria).
2. To compare the tumor response and disease control rate according to Response Evaluation Criteria in Solid Tumors (RECIST1.1), modified Response Evaluation Criteria in Solid Tumors (mRECIST) and European Association of Liver Disease (EASL) criteria.
3. To compare the safety.

OTHER OBJECTIVES:

1. To explore the prognostic value of AFP response after treatment.

OUTLINE: This is a multicenter, phase 3, prospective, randomized, controlled trial. Patients are stratified according to

1. ECOG ( 0 vs. 1)
2. Tumor burden

   1. single vs. multiple lesions
   2. tumor size (>8cm vs. ≤8cm)
   3. vascular invasion (yes vs. no)
   4. extrahepatic metastasis (yes vs. no)
3. Alpha fetoprotein(AFP)(≤ 200 ng/mL vs. > 200 ng/mL) Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening). Patients undergo the first conventional transarterial chemoembolization (TACE) within 3-7 days after the first administration of sorafenib. The conventional TACE consists of an injection containing a mixture of chemotherapeutic agents (doxorubicin) and lipiodol followed by embolization with polyvinyl alcohol (PVA) or beads until complete stasis was achieved in the tumor-feeding vessels. Tumor-feeding vessels should be selected/superselected whenever possible. TACE will be repeated "on demand" depending on the radiological response.

ARM II: Patients receive two tablets of sorafenib (200 mg tablets) twice daily (each morning and evening).

MAINTENANCE THERAPY: Standard follow-up evaluations include contrast-enhanced CT scan and laboratory assessment. Laboratory assessment will be performed every 4 weeks. Radiological follow-up (contrast-enhanced CT scan in liver and chest X-ray) will be performed during week 4 and week 8 after initiation of treatment and thereafter every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Prior informed consent
2. Advanced stage HCC/ Barcelona Clinic Liver Cancer(BCLC) C stage
3. Confirmed Diagnosis of HCC:

   1. Cirrhotic subjects: Clinical diagnosis by Asian Pacific Association for the Study of the Liver(AASLD) criteria.
   2. Non-cirrhotic subjects: for subjects without cirrhosis, histological or cytological confirmation is mandatory
   3. Documentation of original biopsy for diagnosis is acceptable
4. Child Pugh class A without ascites or hepatic encephalopathy
5. Eastern Cooperative Oncology Group(ECOG) Performance Status of 0-1
6. At least one uni-dimensional lesion measurable by CT-scan or MRI according to the RECIST, mRECIST and EASL criteria,respectively

   1. single lesion>5cm
   2. 2-3 lesions, at least one lesion>3cm if more than 4 lesions, no limitation of the tumor size, but the sum of size of all tumor lesions should be less than 50% of liver parenchyma.
7. Male or female subjects ≥ 18 years of age
8. Ability to swallow oral medications
9. Life expectancy of at least 12 weeks
10. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial
11. Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to randomization:

    1. Hemoglobin > 9.0 g/dl
    2. Absolute neutrophil count (ANC) >1,500/mm3
    3. Platelet count≥50x109/L
    4. ALB≥28g/L
    5. Total bilirubin < 2 mg/dL
    6. Alanine aminotransferase(ALT) and aspartate aminotransferase(AST) < 5 x upper limit of normal
    7. Blood urea nitrogen(BUN) and creatinine < 1.5 x upper limit of normal
    8. International normalized ratio(INR) < 1.7, or prothrombin time（PT） < 4 seconds above control

Exclusion Criteria:

1. Diffuse HCC or tumor burden ≥50% of liver parenchyma
2. Main portal vein obstruction, vascular invasion in hepatic vein or inferior vena cava
3. Presence of metastasis in biliary tract,brain or bone
4. Poor blood supply for the liver tumor lesions; poor blood supply refers that the tumor lesions fail to show obvious contrast uptake in the arterial phase and washout in venous or late phases by CT scan or MRI
5. Any contraindications for hepatic embolization procedures:

   1. Known hepatofugal blood flow
   2. Known porto-systemic shunt
   3. Renal failure / insufficiency requiring hemo-or peritoneal dialysis
6. Target lesions having previously been treated with local therapy such as resection of HCC, radiofrequency ablation (RFA), percutaneous ethanol injection (PEI)
7. Other molecular target drugs ongoing or completed < 4 weeks prior to the baseline scan
8. Prior transarterial embolization or systemic chemotherapy
9. Any ≥ CTC adverse events(AEs) grade 2 acute toxic effects of any prior local treatment
10. Patients with untreated varices or active bleeding
11. History of cardiac disease:

    1. Congestive heart failure >New York Heart Association (NYHA) class 2
    2. Uncontrolled hypertension
12. Known history of HIV infection
13. Active clinically serious infections (> grade 2 NCI-CTCAE Version 3.0), except for Hepatitis B virus(HBV) and hepatitis C virus(HCV) infection
14. Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study drug
15. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months prior to the first dose of study drug
16. Previous or concurrent cancer that is distinct in primary site or histology from HCC. Any cancer curatively treated >3 years prior to entry is permitted
17. Any contraindication for sorafenib or doxorubicin administration
18. Pregnant or breast-feeding subjects
19. Any disease(within 6 months of randomization)which could affect the evaluation of the study drug
20. Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
21. Major surgery within 4 weeks prior to start of study drug (e.g. thoracolaparotomy is not allowed, but noninvasive surgery, e.g. biopsy, is allowed)
22. Autologous bone marrow transplant or stem cell rescue within 1 year prior to start of study drug
23. History of organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | The final analysis will occur when the expected number of death (173 events) is reached. Up to 2.5 years
  Overall survival (OS) analysis is measured from the time of randomization until death occurred from any cause.

SECONDARY OUTCOMES:
Time to progression | The time to progression will be assessed at the end of the study, up to 2.5 years
  The time to progression is measured from the time of randomization to the radiologically confirmed progression according to mRECIST criteria.
Tumor response | Tumor response will be assessed up to 2.5 years
  Tumor response will be evaluated according to RECIST, mRECIST and EASL criteria, respectively. Tumor response will be presented in the terms of complete response, partial response, stable disease and progression disease.
Adverse events | The adverse events will be assessed up to 2.5 years.
  The terms and grade of adverse events will be presented according to the Common Terminology Criteria for Adverse Events(CTCAE:version 4.0)

OTHER OUTCOMES:
AFP response | The AFP response will be assessed up to 2.5 years.
  The clinical laboratory will use the electrochemiluminescence immunoassay method to determine the value of AFP. (Elecsys Cobas e601, Roche) ΔAFP(%) = [(AFPbaseline-AFPpost-treatment)/ AFPbaseline]×100%; AFP response =ΔAFP(%) > AFP response cutoff point

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD，PhD, Study Chair — Xijing Hospital of Digestive Disease, Fourth Military Medical University; Guohong Han, MD，PhD, Principal Investigator — Department of Liver Disease and Digestive Interventional Radiology, Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Zhao Y, Wang WJ, Guan S, Li HL, Xu RC, Wu JB, Liu JS, Li HP, Bai W, Yin ZX, Fan DM, Zhang ZL, Han GH. Sorafenib combined with transarterial chemoembolization for the treatment of advanced hepatocellular carcinoma: a large-scale multicenter study of 222 patients. Ann Oncol. 2013 Jul;24(7):1786-1792. doi: 10.1093/annonc/mdt072. Epub 2013 Mar 18. PMID 23508822